CLINICAL TRIAL: NCT00880048
Title: A Randomised, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Orvepitant in Subjects With Major Depressive Disorder
Acronym: Orvepitant MDD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: To allow assessment of isolated events of seizure during program
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110833
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder
Keywords: depression; safety; HAMD; QIDS-SR; NK-1 antagonist; efficacy; orvepitant; placebo; MDD; video-rating
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — orvepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- orvepitant 30 mg (Experimental): orvepitant 30 mg (low dose)
  Interventions: Drug: orvepitant
- orvepitant 60 mg (Experimental): orvepitant 60 mg (high dose)
  Interventions: Drug: orvepitant
- Placebo (Placebo Comparator): inactive placebo to match orvepitant 30 mg and 60 mg dosage forms
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: orvepitant — neurokinin-1 antagonist
  Other Names: GW823296
  Arms: orvepitant 30 mg; orvepitant 60 mg
Other: Placebo — Placebo to match orvepitant 30 mg and 60 mg
  Arms: Placebo

SUMMARY:
This is a 6-week, randomised, multicenter, double-blind, placebo controlled, fixed dose parallel group study to assess the efficacy and safety of orvepitant (30 and 60 mg/day) versus placebo in subjects with a diagnosis of a Major Depressive Disorder, whose symptoms are considered moderate or severe.

Following an initial screening visit, subjects fulfilling the study inclusion and exclusion criteria will enter a pre-treatment screening phase to permit evaluation of the laboratory and ECG assessments and to confirm eligibility for inclusion into the study. This screening phase will be a minimum of 7 days, but no longer than 21 days. At the completion of the screening period, eligible subjects will be randomised at the baseline visit to receive either orvepitant 30mg/day, orvepitant 60mg/day or placebo (equal chance of receiving any of the three possible treatments, i.e., a 1:1:1 ratio) for a six-week double-blind treatment phase. Those subjects randomised to receive placebo will receive study medication identical in appearance to that received by subjects assigned to receive orvepitant 30 or 60mg/day.

Efficacy will be assessed via standard depression symptom and severity rating scales or questionaires. The Hamilton Depression Rating Scale (HAM-D) will be used as the primary measure. Secondary efficacy endpoints include the Quick Inventory of Depressive Symptomatology (QIDS-SR) and the Clinical Global Impression- Global Improvement and Severity of Illness Scale (CGI-I and CGI-S, respectively).

Safety will be assessed by monitoring for adverse events (side effects) and through periodic laboratory evaluations (blood tests), vital signs assessments (e.g., blood pressure, heart rate, temperature) and heart function measurements (electrocardiograms, or ECGs).

DETAILED DESCRIPTION:
The purpose of the current study is to test the safety and the anti-depressant effects of orvepitant, an investigational antidepressant. Efficacy will be assessed using standard depression symptom and severity rating scales (questionaires). The Hamilton Depression Rating Scale (HAM-D) will serve as the primary measure of efficacy, and . Secondary efficacy endpoints include the Bech Melancholia Scale (sum of items 1, 2, 7, 8, 10, and 13 of the 17-item HAM-D scale), the Quick Inventory of Depressive Symptomatology (QIDS-SR), the Clinical Global Impression- Global Improvement and Severity of Illness Scale (CGI-I and CGI-S, respectively), the HAM-D anxiety factor score (sum of items 10, 11, 12, 13, 15 and 17), the Cognitive and Physical Function Questionnaire (CPFQ) and a morning sleep questionnaire.

Safety and tolerability will be assessed by monitoring adverse events (AEs or side effects), physical examinations (including vital signs such as blood pressure and heart rate), clinical laboratory assessments (blood tests), electrical recordings of the heart (electrocardiograms or ECG's), the Columbia Suicidality Severity Rating Scale (CSSRS), Sexual Function Questionnaire (SFQ), and weight change.

Blood samples will be taken at different time points to assess blood levels of orvepitant in patients, allowing the relationship between amount of orvepitant in the body and efficacy to be studied.

The primary objective of the study is to evaluate the antidepressant efficacy of orvepitant (30 and 60mg/day) versus placebo (a "sugar pill", with no active ingredients). The secondary objectives include assessing the safety and tolerability of orvepitant, assessing the profile of appearance and disappearance of orvepitant in the body (blood) following administration (i.e., assessing how long the drug remains in the body), and lastly to examine the relationship between blood levels of the drug and efficacy (i..e, the change in HAM-D total score relative to what it was before starting the study medication.

Following an initial screening visit, subjects fulfilling the study entrance criteria will enter a pre-treatment screening phase to permit evaluation of the laboratory and electrocardiogram assessments and to confirm eligibility for inclusion into the study. This screening phase will be a minimum of 7 days, but no longer than 21 days. During the screening period and the treatment phase if the study, if the subject is selected for study entry, subjects will undergo assessments of their depressive symptoms via a face-to-face interview as well as via a video-based system (i.e., live subject interview conducted by an off-site interviewer using a web-based video camera). Upon completion of the screening period, eligible subjects will be randomly assigned at the baseline visit to one of three treatment regimens: orvepitant 30mg/day, orvepitant 60mg/day or placebo for a six-week treatment phase. The chances of receiving each of the three possible treatments will be equal. Orvepitant will be administered as tablets. Those subjects randomised to receive placebo will receive study medication identical in appearance to that received by subjects assigned to receive orvepitant.

During the treatment phase, subjects will be required to return to the clinic at the end of Weeks 1, 2, 4 and 6. In addition, all subjects will be required to return for a follow-up visit 14 days after the last dose of study medication. In addition, all subjects with ongoing adverse events at the 14-day follow-up visit will be required to return for a further follow-up visit 28 days after the last dose of study medication.

Male and female outpatients between the ages of 18 to 64 years inclusive with a primary diagnosis of Major Depressive Disorder will be enrolled into this study. A total of approximately 350 subjects are expected to be enrolled at approximately 30 different study sites in the U.S. and Canada.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have the ability to comprehend the Informed Consent Form.
* Male or female outpatients, aged 18-64, inclusive.
* A primary diagnosis of major depressive disorder, single episode or recurrent.
* Subjects must, in the investigator's opinion and based on the subject's history, have met depression criteria for at least 8 weeks prior to the Screening Visit.
* Subjects with symptom severity considered to be at least moderate to severe by the investigator.
* Women of childbearing potential are only eligible IF they commit to consistent and correct use of an acceptable method of birth control that must be documentation at each visit

Exclusion Criteria:

* Subjects whose mood-related symptoms are better accounted for by a diagnosis other than depression; subjects diagnosed with Alzheimer's Disease or other form of dementia; subjects diagnosed with a current/recent eating disorder such as anorexia nervosa or bulimia; subjects with a diagnosed history of schizophrenia, schizoaffective disorder, or Bipolar Disorder.
* Subjects with any history of a significant abnormality of the neurological system (including dementia and other cognitive disorders or significant head injury) or any history of seizures (convulsions).
* Subjects have a positive urine test at screening for illegal drug use and/or who have a history of substance abuse or dependence (alcohol or drugs) within the past 12 months.
* Subjects who are currently receiving regularly scheduled psychotherapy (individual or group), plan to start psychotherapy during the trial or have received regularly scheduled psychotherapy during the 12 week period prior to the Screening Visit.
* Subjects who have a history of failing to respond to adequate treatment with an antidepressant, i..e, failure to improve following administration of at least two other antidepressants, each given for at least 4 weeks.
* Subjects who, in the investigator's judgement, pose a homicidal or serious suicidal risk, have made a suicide attempt within the 6 months preceding screening or who have ever been homicidal.
* Subjects who have received the following treatments for depression in the past: electroconvulsive therapy (ECT), vagal stimulation, or transcranial magnetic stimulation (TMS) within the 6 months prior to the Screening Visit.
* Subjects with an unstable medical disorder; or with a disorder that otherwise would likely interfere with the activity of the study medication (orvepitant).
* Subjects have any screening laboratory abnormality that in the investigator's judgement is considered to be clinically significant.
* Subjects with an abnormal thyroid test at the Screening Visit. Subjects maintained on thyroid medication must have normal thyroid levels for a period of at least six months prior to the Screening Visit.
* Subjects have any screening electrocardiography (ECG) finding that in the investigator's judgement is considered to be clinically significant.
* Women who have a positive pregnancy test at the Screening Visit, a positive urine dipstick test at the Baseline (Randomization) Visit, or who are lactating or planning to become pregnant within the 4 months following the Screen Visit.
* Subjects who have taken other psychoactive drugs within two weeks prior to the Baseline Visit i.e. at any time during the Screening period. This includes "over-the-counter" psychoactive medications such as St. John's Wort and SAM-e.
* Subjects who have taken other drugs within 2 weeks prior to the Baseline visit which the investigator feels may interact with the study medication.
* Subjects who are currently participating in another clinical trial in which the subject is or will be exposed to an investigational or non-investigational drug or device, or has done so within the preceding month for studies unrelated to depression, or 6 months for studies related to depression.
* Subjects who have no contact with an adult on a daily basis. This would exclude subjects who are not living with at least one other adult or subjects who do not have an adult who contacts them on a daily basis.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 343 (Actual)
Dates: Start 2009-03-11 (Actual); Primary Completion 2010-06-21 (Actual); Study Completion 2010-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (26):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Weymouth, Massachusetts
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Willingboro, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Garfield Heights, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Salem, Oregon
  - GSK Investigational Site, Emmaus, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Canada (5):
  - GSK Investigational Site, Penticton, British Columbia
  - GSK Investigational Site, Miramichi, New Brunswick
  - GSK Investigational Site, Sydney, Nova Scotia
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Gatineau, Quebec

REFERENCES:
- [Background] Ratti E, Bettica P, Alexander R, Archer G, Carpenter D, Evoniuk G, Gomeni R, Lawson E, Lopez M, Millns H, Rabiner EA, Trist D, Trower M, Zamuner S, Krishnan R, Fava M. Full central neurokinin-1 receptor blockade is required for efficacy in depression: evidence from orvepitant clinical studies. J Psychopharmacol. 2013 May;27(5):424-34. doi: 10.1177/0269881113480990. Epub 2013 Mar 28. PMID 23539641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 centers across the North America (27 centers in United States of America and 4 centers in Canada) during the period 06 April 2009 to 21 June 2010. Total of 1604 participants were screened for study eligibility, of which 343 participants were randomized into the study.
Pre-assignment Details: A total of 339 participants were included in Intent-to-treat (ITT) population. ITT population comprised of all participants who gave informed consent, were randomized, received at least one dose of double blind medication and for whom at least one post-randomization assessment was available.
Groups:
- Placebo: Participants received one tablet of matching placebo, once daily, in the evening for a period of 6 weeks.
- GW823296 30 mg: Participants received one tablet of GW823296 (orvepitant) 30 milligrams (mg), once daily, in the evening for a period of 6 weeks.
- GW823296 60 mg: Participants received one tablet of GW823296 (orvepitant) 60 mg, once daily, in the evening for a period of 6 weeks.
Period: Overall Study
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Started | 116 | 115 | 112
Completed | 88 | 82 | 77
Not Completed | 28 | 33 | 35
Not completed — Adverse Event | 2 | 3 | 5
Not completed — Lack of Efficacy | 1 | 2 | 2
Not completed — Protocol Violation | 4 | 6 | 5
Not completed — Lost to Follow-up | 6 | 6 | 5
Not completed — Physician Decision | 1 | 1 | 7
Not completed — Withdrawal by Subject | 5 | 8 | 5
Not completed — Study closed/terminated | 9 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg | Total
Number analyzed (Participants) | 116 | 115 | 112 | 343
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (10.61) | 40.4 (11.35) | 43.1 (10.66) | 41.7 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 75 | 73 | 216
  Male | 48 | 40 | 39 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 32 | 24 | 33 | 89
  White | 78 | 83 | 76 | 237
  More than one race | 2 | 2 | 2 | 6
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 17-item Hamilton Depression Rating Scale (HAM-D) Total Score
Description: HAM-D was use to measure the severity of depressive symptoms in participants with primary depressive illness. It was a checklist of items that were ranked on a scale of 0-4 or 0-2. Items with quantifiable severity were scored 0 (lowest severity) to 4 (greatest severity); The HAM-D total score was calculated by summing the individual response scores. The lowest possible score was 0 (absence of depression) and the highest possible score was 52 (most severe measure of depression). For the last observation carried forward analyses, the most recent post randomization total score (as opposed to individual responses) was "carried forward" and used in the calculation of the change from randomization (Baseline) value. If the responses to more than 1 question were missing for a participant at a particular time point, the total score was not calculated. Change from Baseline in total score was the difference between HAM-D total score at the time point being analyzed and randomization.
Time Frame: Baseline and up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Scores on a scale
  Week 1: number analyzed (Participants) | 114 | 112 | 107
  Week 1 | -2.85 (0.454) | -4.45 (0.462) | -5.11 (0.470)
  Week 2: number analyzed (Participants) | 107 | 102 | 93
  Week 2 | -4.35 (0.531) | -5.92 (0.545) | -6.00 (0.565)
  Week 4: number analyzed (Participants) | 97 | 92 | 90
  Week 4 | -6.87 (0.672) | -8.68 (0.691) | -8.90 (0.703)
  Week 6: number analyzed (Participants) | 91 | 83 | 76
  Week 6 | -8.29 (0.727) | -9.95 (0.754) | -9.05 (0.777)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 1; Test type: Superiority; p = 0.0133, Mixed Models Repeated Measures; Mean Difference (Net) = -1.60, 95% CI 2-sided [-2.87 to -0.34]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 1; Test type: Superiority; p = 0.0006, Mixed Models Repeated Measures; Mean Difference (Net) = -2.26, 95% CI 2-sided [-3.54 to -0.98]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2; Test type: Superiority; p = 0.0394, Mixed Models Repeated Measures; Mean Difference (Net) = -1.57, 95% CI 2-sided [-3.06 to -0.08]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 2; Test type: Superiority; p = 0.0332, Mixed Models Repeated Measures; Mean Difference (Net) = -1.65, 95% CI 2-sided [-3.16 to -0.13]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 4; Test type: Superiority; p = 0.0601, Mixed Models Repeated Measures; Mean Difference (Net) = -1.82, 95% CI 2-sided [-3.71 to 0.08]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 4; Test type: Superiority; p = 0.0369, Mixed Models Repeated Measures; Mean Difference (Net) = -2.03, 95% CI 2-sided [-3.94 to -0.12]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 6; Test type: Superiority; p = 0.1122, Mixed Models Repeated Measures; Mean Difference (Net) = -1.67, 95% CI 2-sided [-3.73 to 0.39]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 6; Test type: Superiority or Other; p = 0.4713, Mixed Models Repeated Measures; Mean Difference (Net) = -0.76, 95% CI 2-sided [-2.85 to 1.32]

2. Secondary Outcome: Percentage of Participants With a >=50% Reduction From Baseline in HAM-D Total Score
Description: HAM-D was use to measure the severity of depressive symptoms in participants with primary depressive illness. It was a checklist of items that were ranked on a scale of 0-4 or 0-2. The HAM-D Total Score was calculated by summing the individual response scores. The lowest possible score was 0 (absence of depression) and the highest possible score was 52 (most severe measure of depression). For the last observation carried forward analyses, the most recent post randomization total score (as opposed to individual responses) was "carried forward" and used in the calculation of the change from randomization value. If the responses to more than 1 question were missing for a participant at a particular time point, the total score was not calculated. Data was presented as percent of HAM-D responders which was defined as participants who has a >=50% reduction from randomization in HAM-D total score.
Time Frame: Up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Percentage of participants
  Week 1: number analyzed (Participants) | 114 | 112 | 107
  Week 1 | 4 | 7 | 10
  Week 2: number analyzed (Participants) | 107 | 102 | 93
  Week 2 | 9 | 14 | 13
  Week 4: number analyzed (Participants) | 97 | 92 | 90
  Week 4 | 22 | 27 | 29
  Week 6: number analyzed (Participants) | 91 | 83 | 76
  Week 6 | 27 | 37 | 30
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 1; Test type: Superiority; p = 0.2232, Regression, Logistic; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.63 to 7.39]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 1; Test type: Superiority; p = 0.0559, Regression, Logistic; Odds Ratio (OR) = 3.15, 95% CI 2-sided [0.97 to 10.2]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 2; Test type: Superiority; p = 0.3395, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.64 to 3.61]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 2; Test type: Superiority; p = 0.4256, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.59 to 3.50]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 4; Test type: Superiority; p = 0.3790, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.69 to 2.64]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 4; Test type: Superiority; p = 0.2554, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.76 to 2.86]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 6; Test type: Superiority; p = 0.1961, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.80 to 2.91]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 6; Test type: Superiority; p = 0.6916, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.58 to 2.25]

3. Secondary Outcome: Number of Participants Who Maintained Clinical Response by Week 6
Description: The start of the 'maintained antidepressant response' was the time at which a participant demonstrates a 50% reduction from randomization in their HAM-D total score and where this response was maintained until the end of the treatment phase (week 6). Participants who met the 50% reduction at week 6 without having met it at week 4 were considered to have reached a maintained response, and therefore were censored at week 6. Where a participant met the criteria for maintained antidepressant response, the "time (in days) to maintained antidepressant response" was calculated as: (Date of assessment at which the maintained response commences minus Date of randomization) plus 1. Where a participant did not met the criteria for maintained antidepressant response, their time to response was censored at the last on-treatment assessment they undertake, up to and including the week 6 assessment.
Time Frame: Up to Week 6
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Participants | 14 | 20 | 19
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Test type: Superiority; p = 0.61, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.50 to 1.95]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Test type: Superiority; p = 0.35, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.36 to 1.54]

4. Secondary Outcome: Change From Baseline in the Bech Melancholia Scale Total Score (Sum of Items 1, 2, 7, 8, 10, and 13 of the 17-item HAM-D Scale)
Description: The BECH scale was extracted from the HAMD-17 and comprised the 6 items (sum of items 1, 2, 7, 8, 10, and 13 of the 17-item HAM-D scale): Depressed Mood, Feelings of Guilt, Work and Activities, Retardation, Anxiety Psychic and Somatic Symptoms General. The BECH Total Score was calculated by summing the individual response scores. It was a checklist of items that were ranked on a scale of 0-4 or 0-2. The lowest possible score was 0 (absence of depression) and the highest possible score was 22 (most severe measure of depression). Due to the small number of items , missing data was not imputed for the BECH Total Score. If any of the 6 items above were missing, the total score was not calculated at that visit. Value at randomization was the Baseline value. Change from Baseline in BECH Total Score was the difference between BECH Total Score at the time point being analyzed to randomization.
Time Frame: Baseline and up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Scores on a scale
  Week 1: number analyzed (Participants) | 114 | 112 | 107
  Week 1 | -1.24 (0.233) | -1.94 (0.237) | -2.05 (0.241)
  Week 2: number analyzed (Participants) | 107 | 102 | 93
  Week 2 | -2.17 (0.287) | -2.64 (0.296) | -2.79 (0.307)
  Week 4: number analyzed (Participants) | 97 | 92 | 90
  Week 4 | -3.34 (0.357) | -4.01 (0.368) | -4.09 (0.374)
  Week 6: number analyzed (Participants) | 91 | 83 | 76
  Week 6 | -3.69 (0.394) | -4.78 (0.409) | -4.21 (0.421)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 1; Test type: Superiority; p = 0.0362, Mixed Models Repeated Measures; Mean Difference (Net) = -0.69, 95% CI 2-sided [-1.34 to -0.04]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 1; Test type: Superiority; p = 0.0155, Mixed Models Repeated Measures; Mean Difference (Net) = -0.81, 95% CI 2-sided [-1.46 to -0.16]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 2; Test type: Superiority; p = 0.2593, Mixed Models Repeated Measures; Mean Difference (Net) = -0.46, 95% CI 2-sided [-1.27 to 0.34]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 2; Test type: Superiority; p = 0.1407, Mixed Models Repeated Measures; Mean Difference (Net) = -0.62, 95% CI 2-sided [-1.44 to 0.20]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 4; Test type: Superiority; p = 0.1933, Mixed Models Repeated Measures; Mean Difference (Net) = -0.67, 95% CI 2-sided [-1.67 to 0.34]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 4; Test type: Superiority; p = 0.1500, Mixed Models Repeated Measures; Mean Difference (Net) = -0.74, 95% CI 2-sided [-1.76 to 0.27]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 6; Test type: Superiority; p = 0.0550, Mixed Models Repeated Measures; Mean Difference (Net) = -1.09, 95% CI 2-sided [-2.21 to 0.02]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 6; Test type: Superiority; p = 0.3627, Mixed Models Repeated Measures; Mean Difference (Net) = -0.52, 95% CI 2-sided [-1.65 to 0.61]

5. Secondary Outcome: Change From Baseline in the 16-item Quick Inventory of Depressive Symptomatology (QIDS-SR 16) Total Score
Description: QIDS-SR assessed symptoms severity of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criterion for major depressive disorder. It consisted of 16 separate items, defining 9 DSM-IV symptom criterion domains. A total score was obtained by summing scores on each domain. The lowest possible score was 0, which represented an absence of depression; the highest possible score was 27, which represented the most severe measure of depression. Due to the small number of items, missing data was not imputed for the QIDS-SR total score. If any of the 9 domains above were missing, the total score was not calculated at that visit. Value at randomization was the Baseline value. Change from Baseline in total score was the difference between QIDS total score at the time point being analyzed to randomization. If no post- randomization scores were available, change from Baseline was set to missing.
Time Frame: Baseline and up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Scores on a scale
  Week 1: number analyzed (Participants) | 114 | 108 | 107
  Week 1 | -2.14 (0.386) | -3.17 (0.395) | -4.41 (0.399)
  Week 2: number analyzed (Participants) | 106 | 101 | 92
  Week 2 | -3.64 (0.445) | -5.08 (0.455) | -5.48 (0.473)
  Week 4: number analyzed (Participants) | 96 | 92 | 90
  Week 4 | -5.20 (0.498) | -6.78 (0.510) | -7.06 (0.523)
  Week 6: number analyzed (Participants) | 92 | 84 | 74
  Week 6 | -6.17 (0.543) | -7.70 (0.562) | -7.58 (0.588)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 1; Test type: Superiority; p = 0.0616, Mixed Models Repeated Measures; Mean Difference (Net) = -1.03, 95% CI 2-sided [-2.11 to 0.05]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 1; Test type: Superiority; p < 0.0001, Mixed Models Repeated Measures; Mean Difference (Net) = -2.28, 95% CI 2-sided [-3.36 to -1.19]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 2; Test type: Superiority; p = 0.0239, Mixed Models Repeated Measures; Mean Difference (Net) = -1.44, 95% CI 2-sided [-2.68 to -0.19]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 2; Test type: Superiority; p = 0.0048, Mixed Models Repeated Measures; Mean Difference (Net) = -1.84, 95% CI 2-sided [-3.12 to -0.57]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 4; Test type: Superiority; p = 0.0270, Mixed Models Repeated Measures; Mean Difference (Net) = -1.58, 95% CI 2-sided [-2.97 to -0.18]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 4; Test type: Superiority; p = 0.0103, Mixed Models Repeated Measures; Mean Difference (Net) = -1.86, 95% CI 2-sided [-3.27 to -0.44]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 6; Test type: Superiority; p = 0.0497, Mixed Models Repeated Measures; Mean Difference (Net) = -1.53, 95% CI 2-sided [-3.06 to -0.00]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 6; Test type: Superiority; p = 0.0794, Mixed Models Repeated Measures; Mean Difference (Net) = -1.41, 95% CI 2-sided [-2.98 to 0.17]

6. Secondary Outcome: Change From Baseline in the HAM-D Anxiety Factor Score (Sum of Items 10, 11, 12, 13, 15 and 17)
Description: The anxiety score was extracted from the HAM-D-17 and comprises of items 10, 11, 12, 13 and 15 from the HAM-D scale. The anxiety score was calculated by summing the individual response scores to these questions. It was a checklist of items that were ranked on a scale of 0-4 or 0-2. The lowest possible score was 0 (absence of depression) and the highest possible score was 18 (most severe measure of depression). Due to the small number of items, missing data was not imputed for the anxiety score. If either of the anxiety items was missing, the total score was not calculated at that visit. Value at randomization was the Baseline value. Change from Baseline in anxiety score was the difference between the anxiety score at the time point being analyzed to randomization. If no post- randomization scores were available, change from Baseline was set to missing.
Time Frame: Baseline and up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Scores on a scale
  Week 1: number analyzed (Participants) | 114 | 112 | 107
  Week 1 | -0.81 (0.169) | -1.09 (0.172) | -1.57 (0.175)
  Week 2: number analyzed (Participants) | 107 | 102 | 93
  Week 2 | -1.40 (0.185) | -1.55 (0.189) | -1.73 (0.197)
  Week 4: number analyzed (Participants) | 97 | 92 | 90
  Week 4 | -1.96 (0.233) | -2.31 (0.239) | -2.63 (0.243)
  Week 6: number analyzed (Participants) | 91 | 83 | 76
  Week 6 | -2.37 (0.235) | -2.70 (0.244) | -2.56 (0.254)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 1; Test type: Superiority; p = 0.2400, Mixed Models Repeated Measures; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.75 to 0.19]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 1; Test type: Superiority; p = 0.0020, Mixed Models Repeated Measures; Mean Difference (Net) = -0.76, 95% CI 2-sided [-1.23 to -0.28]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 2; Test type: Superiority; p = 0.5605, Mixed Models Repeated Measures; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.67 to 0.36]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 2; Test type: Superiority; p = 0.2215, Mixed Models Repeated Measures; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.86 to 0.20]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 4; Test type: Superiority; p = 0.2870, Mixed Models Repeated Measures; Mean Difference (Net) = -0.35, 95% CI 2-sided [-1.01 to 0.30]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 4; Test type: Superiority; p = 0.0465, Mixed Models Repeated Measures; Mean Difference (Net) = -0.67, 95% CI 2-sided [-1.33 to -0.01]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 6; Test type: Superiority; p = 0.3399, Mixed Models Repeated Measures; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.99 to 0.34]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 6; Test type: Superiority; p = 0.5931, Mixed Models Repeated Measures; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.86 to 0.49]

7. Secondary Outcome: Percentage of Participants With Clinical Global Impression- Global Improvement (CGI-I) Score
Description: The CGI-I assessed scores range from 1 - Very much Improved to 7 - Very much worse, with 0 representing a participant that was not assessed. The assessed scores were dichotomized. Scores of 1 or 2 was in the first category, scoring 1. All other scores (except zero which was regarded as missing) was in the second category, scoring 0. The percentage of participants in the first category was calculated for each assessment.
Time Frame: Up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Percentage of participants
  Week 1: number analyzed (Participants) | 113 | 112 | 108
  Week 1 | 4 | 12 | 9
  Week 2: number analyzed (Participants) | 107 | 101 | 93
  Week 2 | 10 | 25 | 18
  Week 4: number analyzed (Participants) | 97 | 92 | 89
  Week 4 | 33 | 36 | 39
  Week 6: number analyzed (Participants) | 92 | 84 | 76
  Week 6 | 35 | 44 | 42
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 1; Test type: Superiority; p = 0.0562, Regression, Logistic; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.97 to 8.22]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 1; Test type: Superiority; p = 0.1596, Regression, Logistic; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.73 to 6.73]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 2; Test type: Superiority; p = 0.0067, Regression, Logistic; Odds Ratio (OR) = 2.91, 95% CI 2-sided [1.34 to 6.30]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 2; Test type: Superiority; p = 0.1154, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.85 to 4.36]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 4; Test type: Superiority; p = 0.6895, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.62 to 2.07]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 4; Test type: Superiority; p = 0.3654, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.72 to 2.41]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 6; Test type: Superiority; p = 0.2408, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.78 to 2.65]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 6; Test type: Superiority; p = 0.3066, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.74 to 2.60]

8. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Severity of Illness (CGI-S) Score
Description: The CGI-S assessed scores range from 1 - Very much Improved to 7 - Very much worse, with 0 representing a participant that was not assessed. For the CGI-S, remote, blinded MedAvante, raters assessed the participant's severity of illness considering their total clinical experience with the particular population being studied and information obtained during the Baseline HAMD interview with the participant. Value at randomization was the Baseline value. Change from Baseline in total score was the difference between CGI-S Score at the time point being analyzed to randomization. If no post- randomization scores were available, change from Baseline was set to missing.
Time Frame: Baseline and up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Scores on a scale
  Week 1: number analyzed (Participants) | 113 | 112 | 107
  Week 1 | -0.42 (0.075) | -0.57 (0.076) | -0.69 (0.077)
  Week 2: number analyzed (Participants) | 107 | 102 | 93
  Week 2 | -0.58 (0.093) | -0.83 (0.095) | -0.78 (0.099)
  Week 4: number analyzed (Participants) | 97 | 92 | 90
  Week 4 | -0.98 (0.111) | -1.25 (0.114) | -1.26 (0.116)
  Week 6: number analyzed (Participants) | 91 | 83 | 76
  Week 6 | -1.07 (0.123) | -1.45 (0.127) | -1.27 (0.132)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 1; Test type: Superiority; p = 0.1472, Mixed Models Repeated Measures; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.36 to 0.05]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 1; Test type: Superiority; p = 0.0107, Mixed Models Repeated Measures; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.48 to -0.06]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 2; Test type: Superiority; p = 0.0603, Mixed Models Repeated Measures; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.51 to 0.01]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 2; Test type: Superiority; p = 0.1458, Mixed Models Repeated Measures; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.46 to 0.07]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 4; Test type: Superiority; p = 0.0941, Mixed Models Repeated Measures; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.58 to 0.05]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Test type: Superiority; p = 0.0880, Mixed Models Repeated Measures; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.59 to 0.04] — Placebo vs GW823296 60mg: Week 4
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30mg: Week 6; Test type: Superiority; p = 0.0313, Mixed Models Repeated Measures; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.73 to -0.03]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60mg: Week 6; Test type: Superiority; p = 0.2639, Mixed Models Repeated Measures; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.55 to 0.15]

9. Secondary Outcome: Change From Baseline in the Cognitive and Physical Function Questionnaire (CPFQ) Total Score
Description: CPFQ was a brief self-report scale which was designed to measure cognitive and executive dysfunction in mood and anxiety disorders. The CPFQ comprised of 7 questions assessing each of the most common complaints of depressed participants reporting fatigue or cognitive/executive problems. Each question was rated on a scale of 1 to 6, with 1 indicating greater than normal functioning, 2, indicating normal functioning, and with higher numbers indicating poorer functioning. Two versions of the CPFQ were utilized during the study. The Baseline CPFQ requested the participant reflect back over the past month. For the treatment period, the CPFQ requested the participant reflect back over the past week. Value at randomization was the Baseline value. Change from Baseline in Total Score was the difference between CPFQ Score at the time point being analyzed to randomization. If no post- randomization scores were available, change from Baseline was set to missing.
Time Frame: Baseline and up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Scores on a scale
  Week 1: number analyzed (Participants) | 114 | 111 | 107
  Week 1 | -2.56 (0.543) | -4.13 (0.551) | -3.30 (0.560)
  Week 2: number analyzed (Participants) | 107 | 100 | 92
  Week 2 | -3.43 (0.588) | -4.83 (0.605) | -5.37 (0.625)
  Week 4: number analyzed (Participants) | 97 | 89 | 86
  Week 4 | -5.91 (0.631) | -6.68 (0.652) | -6.64 (0.670)
  Week 6: number analyzed (Participants) | 91 | 82 | 75
  Week 6 | -6.34 (0.688) | -7.28 (0.717) | -7.53 (0.746)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1; Test type: Superiority; p = 0.0421, Mixed Models Repeated Measures; Mean Difference (Net) = -1.57, 95% CI 2-sided [-3.08 to -0.06]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1; Test type: Superiority; p = 0.3394, Mixed Models Repeated Measures; Mean Difference (Net) = -0.74, 95% CI 2-sided [-2.27 to 0.78]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2; Test type: Superiority; p = 0.0963, Mixed Models Repeated Measures; Mean Difference (Net) = -1.40, 95% CI 2-sided [-3.05 to 0.25]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2; Test type: Superiority; p = 0.0235, Mixed Models Repeated Measures; Mean Difference (Net) = -1.94, 95% CI 2-sided [-3.62 to -0.26]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4; Test type: Superiority; p = 0.3956, Mixed Models Repeated Measures; Mean Difference (Net) = -0.77, 95% CI 2-sided [-2.54 to 1.01]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4; Test type: Superiority; p = 0.4273, Mixed Models Repeated Measures; Mean Difference (Net) = -0.73, 95% CI 2-sided [-2.53 to 1.07]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6; Test type: Superiority; p = 0.3429, Mixed Models Repeated Measures; Mean Difference (Net) = -0.94, 95% CI 2-sided [-2.89 to 1.01]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6; Test type: Superiority; p = 0.2403, Mixed Models Repeated Measures; Mean Difference (Net) = -1.19, 95% CI 2-sided [-3.18 to 0.80]

10. Secondary Outcome: Change From Baseline in Morning Sleep Questionnaire (MSQ) Total Sleep Time, Sleep Onset Latency and Wake Time After Sleep Onset
Description: The MSQ was a self-rated scale designed to assess effects on sleep and effects on next day functioning. The following variables were assessed in order to determine effects on sleep: total sleep time, sleep onset latency, number of nocturnal awakenings, wake time after sleep onset and sleep quality (from poor, assigned a score of 1, to excellent, assigned a score of 10). The refreshing value of the sleep was also determined (poor assigned a score of 1, to excellent, assigned a score of 10). Value at randomization was the Baseline value. Change from Baseline was calculated for each domain separately. Change from Baseline was the difference between score at the time point being analyzed to randomization. If no post- randomization scores were available, change from Baseline was set to missing.
Time Frame: Baseline and up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: minutes (min)
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
minutes (min)
  Week 1, total sleep time: number analyzed (Participants) | 111 | 109 | 104
  Week 1, total sleep time | 20.79 (9.733) | 43.31 (9.800) | 54.00 (10.056)
  Week 2, total sleep time: number analyzed (Participants) | 103 | 101 | 94
  Week 2, total sleep time | 34.02 (9.635) | 41.64 (9.743) | 55.42 (10.128)
  Week 4, total sleep time: number analyzed (Participants) | 97 | 90 | 89
  Week 4, total sleep time | 33.07 (10.144) | 63.94 (10.463) | 69.59 (10.641)
  Week 6, total sleep time: number analyzed (Participants) | 90 | 81 | 73
  Week 6, total sleep time | 52.03 (9.986) | 54.21 (10.394) | 80.43 (10.956)
  Week 1, sleep onset latency: number analyzed (Participants) | 111 | 109 | 104
  Week 1, sleep onset latency | -12.50 (6.310) | -36.40 (6.372) | -37.99 (6.547)
  Week 2, sleep onset latency: number analyzed (Participants) | 103 | 101 | 94
  Week 2, sleep onset latency | -21.70 (7.417) | -34.15 (7.508) | -19.95 (7.815)
  Week 4, sleep onset latency: number analyzed (Participants) | 97 | 90 | 89
  Week 4, sleep onset latency | -27.84 (6.940) | -40.76 (7.143) | -38.39 (7.290)
  Week 6, sleep onset latency: number analyzed (Participants) | 90 | 81 | 73
  Week 6, sleep onset latency | -18.93 (8.284) | -47.51 (8.684) | -48.99 (9.163)
  Week 1, wake time after sleep onset: number analyzed (Participants) | 85 | 81 | 74
  Week 1, wake time after sleep onset | 4.61 (4.661) | -12.58 (4.807) | -11.54 (5.061)
  Week 2, wake time after sleep onset: number analyzed (Participants) | 83 | 73 | 68
  Week 2, wake time after sleep onset | -8.10 (5.652) | -6.21 (6.061) | -2.83 (6.298)
  Week 4, wake time after sleep onset: number analyzed (Participants) | 70 | 60 | 57
  Week 4, wake time after sleep onset | -7.36 (5.087) | -9.86 (5.505) | -16.80 (5.670)
  Week 6, wake time after sleep onset: number analyzed (Participants) | 61 | 52 | 46
  Week 6, wake time after sleep onset | 1.34 (6.926) | -13.17 (7.479) | -15.76 (7.932)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1, total sleep time; Test type: Superiority; p = 0.1030, Mixed Models Repeated Measures; Mixed effects repeated measures model = 22.52, 95% CI 2-sided [-4.58 to 49.61]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1, total sleep time; Test type: Superiority; p = 0.0179, Mixed Models Repeated Measures; Mean Difference (Net) = 33.21, 95% CI 2-sided [5.76 to 60.65]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2, total sleep time; Test type: Superiority; p = 0.5773, Mixed Models Repeated Measures; Mean Difference (Net) = 7.62, 95% CI 2-sided [-19.25 to 34.49]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2, total sleep time; Test type: Superiority; p = 0.1250, Mixed Models Repeated Measures; Mean Difference (Net) = 21.40, 95% CI 2-sided [-5.97 to 48.76]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4, total sleep time; Test type: Superiority; p = 0.0344, Mixed Models Repeated Measures; Mean Difference (Net) = 30.87, 95% CI 2-sided [2.29 to 59.45]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4, total sleep time; Test type: Superiority; p = 0.0131, Mixed Models Repeated Measures; Mean Difference (Net) = 36.52, 95% CI 2-sided [7.72 to 65.32]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6, total sleep time; Test type: Superiority; p = 0.8794, Mixed Models Repeated Measures; Mean Difference (Net) = 2.18, 95% CI 2-sided [-26.10 to 30.46]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6, total sleep time; Test type: Superiority; p = 0.0556, Mixed Models Repeated Measures; Mean Difference (Net) = 28.40, 95% CI 2-sided [-0.69 to 57.50]
Statistical Analysis 9: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1, sleep onset latency; Test type: Superiority; p = 0.0078, Mixed Models Repeated Measures; Mean Difference (Net) = -23.90, 95% CI 2-sided [-41.46 to -6.33]
Statistical Analysis 10: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1, sleep onset latency; Test type: Superiority; p = 0.0052, Mixed Models Repeated Measures; Mean Difference (Net) = -25.49, 95% CI 2-sided [-43.30 to -7.68]
Statistical Analysis 11: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2, sleep onset latency; Test type: Superiority; p = 0.2373, Mixed Models Repeated Measures; Mean Difference (Net) = -12.45, 95% CI 2-sided [-33.14 to 8.24]
Statistical Analysis 12: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2, sleep onset latency; Test type: Superiority; p = 0.8707, Mixed Models Repeated Measures; Mean Difference (Net) = 1.75, 95% CI 2-sided [-19.38 to 22.87]
Statistical Analysis 13: Comparison: Placebo vs GW823296 30 mg; Placebo va GW823296 30 mg: Week 4, sleep onset latency; Test type: Superiority; p = 0.1933, Mixed Models Repeated Measures; Mean Difference (Net) = -12.92, 95% CI 2-sided [-32.43 to 6.59]
Statistical Analysis 14: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4, sleep onset latency; Test type: Superiority; p = 0.2933, Mixed Models Repeated Measures; Mean Difference (Net) = -10.55, 95% CI 2-sided [-30.26 to 9.17]
Statistical Analysis 15: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6, sleep onset latency; Test type: Superiority; p = 0.0177, Mixed Models Repeated Measures; Mean Difference (Net) = -28.58, 95% CI 2-sided [-52.15 to -5.01]
Statistical Analysis 16: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6, sleep onset latency; Test type: Superiority; p = 0.0152, Mixed Models Repeated Measures; Mean Difference (Net) = -30.07, 95% CI 2-sided [-54.29 to -5.84]
Statistical Analysis 17: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1, wake time after sleep onset; Test type: Superiority; p = 0.0108, Mixed Models Repeated Measures; Mean Difference (Net) = -17.19, 95% CI 2-sided [-30.36 to -4.01]
Statistical Analysis 18: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1, wake time after sleep onset; Test type: Superiority; p = 0.0190, Mixed Models Repeated Measures; Mean Difference (Net) = -16.15, 95% CI 2-sided [-29.61 to -2.68]
Statistical Analysis 19: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2, wake time after sleep onset; Test type: Superiority; p = 0.8195, Mixed Models Repeated Measures; Mean Difference (Net) = 1.89, 95% CI 2-sided [-14.43 to 18.21]
Statistical Analysis 20: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2, wake time after sleep onset; Test type: Superiority; p = 0.5327, Mixed Models Repeated Measures; Mean Difference (Net) = 5.27, 95% CI 2-sided [-11.35 to 21.89]
Statistical Analysis 21: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4, wake time after sleep onset; Test type: Superiority; p = 0.7387, Mixed Models Repeated Measures; Mean Difference (Net) = -2.50, 95% CI 2-sided [-17.24 to 12.25]
Statistical Analysis 22: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4, wake time after sleep onset; Test type: Superiority; p = 0.2134, Mixed Models Repeated Measures; Mean Difference (Net) = -9.44, 95% CI 2-sided [-24.35 to 5.48]
Statistical Analysis 23: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6, wake time after sleep onset; Test type: Superiority; p = 0.1561, Mixed Models Repeated Measures; Mean Difference (Net) = -14.51, 95% CI 2-sided [-34.61 to 5.60]
Statistical Analysis 24: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6, wake time after sleep onset; Test type: Superiority; p = 0.1054, Mixed Models Repeated Measures; Mean Difference (Net) = -17.10, 95% CI 2-sided [-37.84 to 3.64]

11. Secondary Outcome: Change From Baseline in the MSQ Number of Nocturnal Awakenings
Description: as for outcome 10
Time Frame: Baseline and upto Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Number of awakenings
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Number of awakenings
  Week 1: number analyzed (Participants) | 85 | 81 | 74
  Week 1 | -0.06 (0.130) | -0.63 (0.134) | -0.16 (0.141)
  Week 2: number analyzed (Participants) | 83 | 73 | 68
  Week 2 | -0.52 (0.116) | -0.77 (0.124) | -0.47 (0.130)
  Week 4: number analyzed (Participants) | 70 | 60 | 57
  Week 4 | -0.38 (0.174) | -0.43 (0.187) | -0.78 (0.194)
  Week 6: number analyzed (Participants) | 61 | 52 | 46
  Week 6 | -0.63 (0.152) | -0.42 (0.165) | -0.87 (0.175)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1; Test type: Superiority; p = 0.0024, Mixed Models Repeated Measures; Mean Difference (Net) = -0.57, 95% CI 2-sided [-0.94 to -0.21]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1; Test type: Superiority; p = 0.6146, Mixed Models Repeated Measures; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.47 to 0.28]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2; Test type: Superiority; p = 0.1442, Mixed Models Repeated Measures; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.59 to 0.09]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2; Test type: Superiority; p = 0.8001, Mixed Models Repeated Measures; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.30 to 0.39]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4; Test type: Superiority; p = 0.8439, Mixed Models Repeated Measures; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.55 to 0.45]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4; Test type: Superiority; p = 0.1259, Mixed Models Repeated Measures; Mean Difference (Net) = -0.40, 95% CI 2-sided [-0.91 to 0.11]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6; Test type: Superiority; p = 0.3709, Mixed Models Repeated Measures; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.24 to 0.64]
Statistical Analysis 8: Comparison: Placebo; Placebo vs GW823296 60 mg: Week 6; Test type: Superiority; p = 0.2993, Mixed Models Repeated Measures; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.70 to 0.22]

12. Secondary Outcome: Change From Baseline in the MSQ Sleep Quality and Refreshing Value of Sleep
Description: as for outcome 10
Time Frame: Baseline and up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Scores on a scale
  Week 1, sleep quality: number analyzed (Participants) | 111 | 109 | 104
  Week 1, sleep quality | 0.73 (0.196) | 1.32 (0.198) | 1.45 (0.203)
  Week 2, sleep quality: number analyzed (Participants) | 103 | 101 | 94
  Week 2, sleep quality | 1.03 (0.204) | 1.46 (0.206) | 1.54 (0.214)
  Week 4, sleep quality: number analyzed (Participants) | 97 | 90 | 89
  Week 4, sleep quality | 1.39 (0.212) | 2.12 (0.219) | 1.82 (0.222)
  Week 6, sleep quality: number analyzed (Participants) | 90 | 81 | 73
  Week 6, sleep quality | 1.77 (0.234) | 2.34 (0.243) | 2.09 (0.254)
  Week 1, refreshing value of sleep: number analyzed (Participants) | 111 | 109 | 104
  Week 1, refreshing value of sleep | 0.97 (0.193) | 1.31 (0.195) | 1.60 (0.200)
  Week 2, refreshing value of sleep: number analyzed (Participants) | 103 | 101 | 94
  Week 2, refreshing value of sleep | 1.15 (0.201) | 1.48 (0.203) | 1.80 (0.211)
  Week 4, refreshing value of sleep: number analyzed (Participants) | 97 | 90 | 89
  Week 4, refreshing value of sleep | 1.61 (0.216) | 2.30 (0.223) | 2.00 (0.227)
  Week 6, refreshing value of sleep: number analyzed (Participants) | 90 | 81 | 73
  Week 6, refreshing value of sleep | 1.86 (0.242) | 2.23 (0.252) | 2.57 (0.264)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1, sleep quality; Test type: Superiority; p = 0.0344, Mixed Models Repeated Measures; Mean Difference (Net) = 0.59, 95% CI 2-sided [0.04 to 1.14]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1, sleep quality; Test type: Superiority; p = 0.0111, Mixed Models Repeated Measures; Mean Difference (Net) = 0.72, 95% CI 2-sided [0.17 to 1.27]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2, sleep quality; Test type: Superiority; p = 0.1443, Mixed Models Repeated Measures; Mean Difference (Net) = 0.42, 95% CI 2-sided [-0.15 to 0.99]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2, sleep quality; Test type: Superiority; p = 0.0873, Mixed Models Repeated Measures; Mean Difference (Net) = 0.50, 95% CI 2-sided [-0.07 to 1.08]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4, sleep quality; Test type: Superiority; p = 0.0170, Mixed Models Repeated Measures; Mean Difference (Net) = 0.73, 95% CI 2-sided [0.13 to 1.33]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4, sleep quality; Test type: Superiority; p = 0.1675, Mixed Models Repeated Measures; Mean Difference (Net) = 0.42, 95% CI 2-sided [-0.18 to 1.02]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6, sleep quality; Test type: Superiority; p = 0.0956, Mixed Models Repeated Measures; Mean Difference (Net) = 0.56, 95% CI 2-sided [-0.10 to 1.23]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6, sleep quality; Test type: Superiority; p = 0.3503, Mixed Models Repeated Measures; Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.35 to 1.00]
Statistical Analysis 9: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1, refreshing value of sleep; Test type: Superiority; p = 0.2147, Mixed Models Repeated Measures; Mean Difference (Net) = 0.34, 95% CI 2-sided [-0.20 to 0.88]
Statistical Analysis 10: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1, refreshing value of sleep; Test type: Superiority; p = 0.0233, Mixed Models Repeated Measures; Mean Difference (Net) = 0.63, 95% CI 2-sided [0.09 to 1.17]
Statistical Analysis 11: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2, refreshing value of sleep; Test type: Superiority; p = 0.2404, Mixed Models Repeated Measures; Mean Difference (Net) = 0.33, 95% CI 2-sided [-0.22 to 0.89]
Statistical Analysis 12: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2, refreshing value of sleep; Test type: Superiority; p = 0.0247, Mixed Models Repeated Measures; Mean Difference (Net) = 0.65, 95% CI 2-sided [0.08 to 1.22]
Statistical Analysis 13: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4, refreshing value of sleep; Test type: Superiority; p = 0.0271, Mixed Models Repeated Measures; Mean Difference (Net) = 0.69, 95% CI 2-sided [0.08 to 1.29]
Statistical Analysis 14: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4, refreshing value of sleep; Test type: Superiority; p = 0.2129, Mixed Models Repeated Measures; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.22 to 1.00]
Statistical Analysis 15: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6, refreshing value of sleep; Test type: Superiority; p = 0.2874, Mixed Models Repeated Measures; Mean Difference (Net) = 0.37, 95% CI 2-sided [-0.31 to 1.06]
Statistical Analysis 16: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6, refreshing value of sleep; Test type: Superiority; p = 0.0472, Mixed Models Repeated Measures; Mean Difference (Net) = 0.71, 95% CI 2-sided [0.01 to 1.41]

13. Secondary Outcome: Number of HAM-D Remitters
Description: A HAMD remitter was defined as a participant who had a HAMD Total Score <=7. The HAMD total score was calculated for each participant at each time point. Those participants with no missing value for HAMD total score were categorized as having a HAMD total score of <=7 or >7.
Time Frame: Up to Week 6
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 112 | 111
Participants
  Week 1: number analyzed (Participants) | 114 | 112 | 107
  Week 1 | 2 | 2 | 1
  Week 2: number analyzed (Participants) | 107 | 102 | 93
  Week 2 | 3 | 3 | 5
  Week 4: number analyzed (Participants) | 97 | 92 | 90
  Week 4 | 6 | 13 | 14
  Week 6: number analyzed (Participants) | 91 | 83 | 76
  Week 6 | 10 | 19 | 11
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1; Test type: Superiority; p = 0.9824, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.13 to 7.09]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1; Test type: Superiority; p = 0.6227, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.05 to 6.13]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2; Test type: Superiority; p = 0.9967, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.20 to 5.07]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2; Test type: Superiority; p = 0.3550, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.46 to 8.63]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4; Test type: Superiority; p = 0.1009, Regression, Logistic; Odds Ratio (OR) = 2.35, 95% CI 2-sided [0.85 to 6.49]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4; Test type: Superiority; p = 0.0455, Regression, Logistic; Odds Ratio (OR) = 2.80, 95% CI 2-sided [1.02 to 7.68]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6; Test type: Superiority; p = 0.0507, Regression, Logistic; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.00 to 5.32]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6; Test type: Superiority; p = 0.4962, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.55 to 3.45]

14. Secondary Outcome: Number of Participants With Suicide-Related Events Based on the Columbia Suicidality Severity Rating Scale (CSSRS)
Description: Assessment of suicidality were done through use of the CSSRS for suicidal ideation and suicidal behavior. For suicidal ideation ratings were 1 to 5, where 1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation without intent to act, 4. Active suicidal ideation with any methods (not plan) without intent to act, 5. Active suicidal ideation with specific plan and intent and for suicidal behavior ratings were 6 to 12, Where 6. Actual attempt, 7. Engaged in non-suicidal self-injurious behavior, 8. Interrupted attempt, 9. Aborted attempt, 10. Preparatory acts or behavior, 11. Suicidal behavior, 12. Completed suicide. n= number participants with at least one CSSRS assessment after the first dose of study medication (i.e. on treatment or post treatment). Only those categories from CSSRS (1-12) are presented for which symptoms were actually observed in the participants. Categories with null values for all the arms have not been presented.
Time Frame: Up to 17 days post-treatment
Population: The All Subjects Population was defined as all participants who received at least one dose of study medication. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 115 | 112 | 111
Participants
  Wish to be dead | 46 | 41 | 36
  Non-specific active suicidal thoughts | 12 | 12 | 11
  Active SI without intent to act (ITA) | 8 | 9 | 6
  Active SI with any methods (not plan) without ITA | 1 | 2 | 0
  Active SI with specific plan and intent | 0 | 1 | 0
  Engaged in non-suicidal self-injurious behavior | 1 | 0 | 0

15. Secondary Outcome: Number of Incidences of Discontinuation Emergent Signs and Symptoms Using the Discontinuation-Emergent Signs and Symptoms (DESS)
Description: The DESS scale consisted of 43 signs and symptoms, scored as 'new symptom', 'old symptom but worse', 'old symptom but improved' or 'symptom not present/old symptom but unchanged'. The total number of new signs and symptoms, old symptoms but worse, old symptoms but improved and the total number of new or old-but-worse signs and symptoms were calculated for each treatment and visit. n = number of subjects who had at least one of the 43 symptoms in the specified category. The summary for a specified category are of the number of symptoms the n subjects had in that category. Treatment period was up to Week 6.
Time Frame: Up to 17 days post-treatment
Population: All subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Number of Incidences
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 116 | 115 | 112
Number of Incidences
  New Symptom: number analyzed (Participants) | 0 | 2 | 3
  New Symptom |  | 6.0 (5.66) | 2.7 (1.53)
  Old Symptom But Improved: number analyzed (Participants) | 1 | 2 | 2
  Old Symptom But Improved | 1.0 (NA) — Only one participant was analyzed | 5.0 (5.66) | 3.0 (1.41)
  Old Symptom But Worsened: number analyzed (Participants) | 0 | 2 | 4
  Old Symptom But Worsened |  | 7.5 (0.71) | 4.3 (3.77)
  Unchanged/ Not present: number analyzed (Participants) | 3 | 4 | 9
  Unchanged/ Not present | 42.7 (0.58) | 33.8 (6.60) | 39.6 (5.34)
  New or Old but Worsened: number analyzed (Participants) | 0 | 3 | 5
  New or Old but Worsened |  | 9.0 (7.55) | 5.0 (4.30)

16. Secondary Outcome: Change From Baseline in the Massachusetts Sexual Function Questionnaire (MSFQ) Total Score in Males
Description: MSFQ included five items with a score ranging from 1 to 6 (1 = greater than normal; 2 = normal; 3 = minimally diminished; 5 = markedly diminished; and 6 = totally absent). The following areas of sexual functioning were included: diminished/absent libido; arousal difficulties; orgasm difficulties/anorgasmia; erectile dysfunction (males only) and degree of sexual satisfaction. A total score was used as a global measure of sexual dysfunction. The Baseline MSFQ requested the participant reflect back over the past month. For the treatment period, the follow-up MSFQ requested the participant reflect back over the past week. Change from Baseline was the value at post-Baseline visit minus Baseline value.
Time Frame: Baseline and up to Week 6
Population: All subjects Population (males). Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 48 | 40 | 39
Scores on a scale
  Week 1: number analyzed (Participants) | 46 | 38 | 37
  Week 1 | -1.88 (0.690) | -0.84 (0.787) | -2.43 (0.795)
  Week 2: number analyzed (Participants) | 43 | 33 | 31
  Week 2 | -3.44 (0.840) | -1.00 (0.968) | -2.53 (0.988)
  Week 4: number analyzed (Participants) | 36 | 30 | 29
  Week 4 | -3.88 (1.003) | -3.70 (1.122) | -4.59 (1.141)
  Week 6: number analyzed (Participants) | 34 | 27 | 23
  Week 6 | -3.79 (1.136) | -4.47 (1.269) | -4.46 (1.322)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1; Test type: Superiority; p = 0.3241, Mixed Models Repeated Measures; Mean Difference (Net) = 1.03, 95% CI 2-sided [-1.03 to 3.10]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1; Test type: Superiority; p = 0.6020, Mixed Models Repeated Measures; Mean Difference (Net) = -0.56, 95% CI 2-sided [-2.66 to 1.55]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2; Test type: Superiority; p = 0.0594, Mixed Models Repeated Measures; Mean Difference (Net) = 2.44, 95% CI 2-sided [-0.10 to 4.99]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2; Test type: Superiority; p = 0.4828, Mixed Models Repeated Measures; Mean Difference (Net) = 0.92, 95% CI 2-sided [-1.67 to 3.50]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4; Test type: Superiority; p = 0.9008, Mixed Models Repeated Measures; Mean Difference (Net) = 0.19, 95% CI 2-sided [-2.80 to 3.18]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4; Test type: Superiority; p = 0.6428, Mixed Models Repeated Measures; Mean Difference (Net) = -0.71, 95% CI 2-sided [-3.74 to 2.32]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6; Test type: Superiority; p = 0.6911, Mixed Models Repeated Measures; Mean Difference (Net) = -0.68, 95% CI 2-sided [-4.06 to 2.70]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6; Test type: Superiority; p = 0.7026, Mixed Models Repeated Measures; Odds Ratio (OR) = -0.67, 95% CI 2-sided [-4.14 to 2.80]

17. Secondary Outcome: Change From Baseline in the MSFQ Total Score in Females
Description: as for outcome 16
Time Frame: Baseline and up to Week 6
Population: All Subject Population (female). Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
Number analyzed (Participants) | 68 | 75 | 73
scores on a scale
  Week 1: number analyzed (Participants) | 68 | 72 | 71
  Week 1 | 0.15 (0.473) | -0.82 (0.473) | 0.62 (0.467)
  Week 2: number analyzed (Participants) | 64 | 65 | 62
  Week 2 | -0.62 (0.577) | -1.38 (0.578) | 0.32 (0.578)
  Week 4: number analyzed (Participants) | 61 | 59 | 61
  Week 4 | -1.64 (0.645) | -2.62 (0.653) | -1.58 (0.645)
  Week 6: number analyzed (Participants) | 57 | 54 | 52
  Week 6 | -2.39 (0.699) | -2.94 (0.718) | -1.68 (0.724)
Statistical Analysis 1: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 1; Test type: Superiority; p = 0.1301, Mixed Models Repeated Measures; Mean Difference (Net) = -0.97, 95% CI 2-sided [-2.24 to 0.29]
Statistical Analysis 2: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 1; Test type: Superiority; p = 0.4644, Mixed Models Repeated Measures; Mean Difference (Net) = 0.47, 95% CI 2-sided [-0.79 to 1.73]
Statistical Analysis 3: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 2; Test type: Superiority; p = 0.3382, Mixed Models Repeated Measures; Mean Difference (Net) = -0.76, 95% CI 2-sided [-2.33 to 0.80]
Statistical Analysis 4: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 2; Test type: Superiority; p = 0.2410, Mixed Models Repeated Measures; Mean Difference (Net) = 0.94, 95% CI 2-sided [-0.63 to 2.51]
Statistical Analysis 5: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 4; Test type: Superiority; p = 0.2768, Mixed Models Repeated Measures; Mean Difference (Net) = -0.98, 95% CI 2-sided [-2.75 to 0.79]
Statistical Analysis 6: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 4; Test type: Superiority; p = 0.9434, Mixed Models Repeated Measures; Mean Difference (Net) = 0.06, 95% CI 2-sided [-1.70 to 1.83]
Statistical Analysis 7: Comparison: Placebo vs GW823296 30 mg; Placebo vs GW823296 30 mg: Week 6; Test type: Superiority; p = 0.5796, Mixed Models Repeated Measures; Mean Difference (Net) = -0.55, 95% CI 2-sided [-2.49 to 1.40]
Statistical Analysis 8: Comparison: Placebo vs GW823296 60 mg; Placebo vs GW823296 60 mg: Week 6; Test type: Superiority; p = 0.4753, Mixed Models Repeated Measures; Mean Difference (Net) = 0.71, 95% CI 2-sided [-1.24 to 2.66]

ADVERSE EVENTS:
Time Frame: AEs were reported up to follow up (28 day) post-treatment (Week 6)
Description: AEs were reported for the All subjects Population which was defined as all participants who received at least one dose of study medication.
Arm/Group | Placebo | GW823296 30 mg | GW823296 60 mg
All-Cause Mortality (participants affected / at risk) | 1/116 | 0/115 | 0/112
Serious Adverse Events (participants affected / at risk) | 1/116 | 1/115 | 3/112
Other Adverse Events (participants affected / at risk) | 52/116 | 61/115 | 62/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=116) | GW823296 30 mg (N=115) | GW823296 60 mg (N=112)
Convulsion (Nervous system disorders) | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=116) | GW823296 30 mg (N=115) | GW823296 60 mg (N=112)
Dry mouth (Gastrointestinal disorders) | 14 | 11 | 12
Nausea (Gastrointestinal disorders) | 16 | 8 | 10
Diarrhoea (Gastrointestinal disorders) | 8 | 12 | 10
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 6
Flatulence (Gastrointestinal disorders) | 6 | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 7
Headache (Nervous system disorders) | 19 | 19 | 24
Somnolence (Nervous system disorders) | 6 | 12 | 8
Dizziness (Nervous system disorders) | 4 | 9 | 8
Insomnia (Psychiatric disorders) | 2 | 4 | 9
Anxiety (Psychiatric disorders) | 2 | 6 | 5
Fatigue (General disorders) | 2 | 9 | 7
Upper respiratory tract infection (Infections and infestations) | 4 | 7 | 7

LIMITATIONS AND CAVEATS:
The study was terminated early upon the recommendation of an Independent Data Monitoring Committee. At the time the trial was terminated 343 participants had been randomized, compared to a target of 348 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.